CLINICAL TRIAL: NCT03737942
Title: Effect of Type II Diabetes Mellitus With Neuropathy on the Clinical Use of Rocuronium: A Pharmacodynamic Modelling Study
Brief Title: Effect of Type II Diabetes Mellitus With Neuropathy on the Clinical Use of Rocuronium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, principal investigator, Assiut University
Other Study IDs: Type II DM with Neuropathy
Record Dates: First submitted 2018-11-04; First posted 2018-11-13 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Neuromuscular Transmission Disorder; Diabetes Mellitus, Type 2
Keywords: diabetes mellitus; Neuromuscular Transmission
MeSH Terms: conditions — Neuromuscular Junction Diseases; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group: Motor nerve conduction studies:
  Were done on right ulner, right median, right common peroneal, and right anterior tibial nerves F-wave (for Median, Ulnar and common peroneal nerves) H-reflex study
  Interventions: Device: monitoring of neuromuscular function
- T2DM without neuropathy: Motor nerve conduction studies:
  Were done on right ulner, right median, right common peroneal, and right anterior tibial nerves F-wave (for Median, Ulnar and common peroneal nerves) H-reflex study
  Interventions: Device: monitoring of neuromuscular function
- T2DM with neuropathy: Motor nerve conduction studies:
  Were done on right ulner, right median, right common peroneal, and right anterior tibial nerves F-wave (for Median, Ulnar and common peroneal nerves) H-reflex study
  Interventions: Device: monitoring of neuromuscular function

INTERVENTIONS:
Device: monitoring of neuromuscular function — started by percutaneous stimulation of the cubital nerve at the wrist level
  Other Names: acceleromyographic device

SUMMARY:
International Diabetes Federation estimates that there are now 415 million adults aged 20-79 with diabetes mellitus worldwide. By 2040 this will rise to 640 million. Although diabetes mellitus is highly prevalent in our environment and one of the most important challenges of modern medicine, only a handful of studies have examined the neuromuscular function in diabetic patients. The shortage of publications in this area is still more surprising if we consider that the neuromuscular blockers are one of the pillars in the administration of general anesthesia. Neuromuscular blockers during surgery are used in tracheal intubation and to improve surgical conditions.

DETAILED DESCRIPTION:
In diabetic patients, neuropathy, microvascular and macrovascular complications are known clinical findings which require attention during anesthesia. Partial degeneration or segmental demyelination of the nerve fibers and loss of motor units have been reported in patients with diabetes mellitus as well. Therefore, the effects of a neuromuscular blocking agent should be important because of potential complications from incomplete reversal or residual paralysis during anesthesia maintenance. In a series of studies, vecuronium has been the only agent investigated in patients with diabetes mellitus and other diseases characterized by neuromuscular dysfunction. Delayed recovery from the neuromuscular block after vecuronium administration was shown in patients with diabetes mellitus. Currently, rocuronium, with its rapid onset of action, rapid recovery profile and inactive metabolites, is generally known as a safe agent for anesthesia under normal conditions. It is known that the pharmacokinetic properties of rocuronium can be altered in some diseases, such as renal or hepatic failure. However, it has not been investigated whether the effect of rocuronium on neuromuscular function is changed in the presence of neuropathy in diabetes mellitus patients or not. The rationale of our study arises from the finding of many studies that show different changes in the neurophysiological parameters in diabetes mellitus. In diabetic nerve, the conduction velocity of the action potential is decreased, the amplitude of action potentials, both sensory and motor, is smaller, and the latency time is elongated.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged from 18 years to 65 years.
* scheduled for abdominal surgery under general anesthesia

Exclusion Criteria:

* Patients with allergy to rocuronium
* those diagnosed with diseases that alter neuromuscular blocker response (e.g., Guillain-Barré syndrome, Duchenne type muscle dystrophies, etc.),
* patients receiving treatment with drugs capable of altering neuromuscular transmission or neuromuscular blocker response (e.g., antiseizure drugs, certain antibiotics, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * patients with diabetes Mellitus type 2.
  * Patients with suspected difficult airway (Mallampati class III and IV, thyromental distance <6.5 cm, oral aperture <3.5 cm) were also excluded.
  * In relation to kidney function, patients with serum creatinine ≥1.5 mg/dl or more were excluded.
  * we excluded individuals with GPT or GOT enzyme values ≥42 IU/l or a body mass index (BMI) of <18.5 kg/m2 or > 30 kg/m2.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-01-15 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
neuromuscular monitoring | before operation,till one hour
  Tetanic stimulus , 50 Hz during 5 seconds (tetanic preconditioning).

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Abo Elfadl, M.D, Principal Investigator — Assiut University
Locations (1):
- Assiut governorate, Asyut, Egypt

REFERENCES:
- [Background] Hafeez KR, Tuteja A, Singh M, Wong DT, Nagappa M, Chung F, Wong J. Postoperative complications with neuromuscular blocking drugs and/or reversal agents in obstructive sleep apnea patients: a systematic review. BMC Anesthesiol. 2018 Jul 19;18(1):91. doi: 10.1186/s12871-018-0549-x. PMID 30025517
- [Background] Nandi R, Basu SR, Sarkar S, Garg R. A comparison of haemodynamic responses between clinical assessment-guided tracheal intubation and neuromuscular block monitoring-guided tracheal intubation: A prospective, randomised study. Indian J Anaesth. 2017 Nov;61(11):910-915. doi: 10.4103/ija.IJA_93_17. PMID 29217857
- [Background] Kashiwai A, Suzuki T, Ogawa S. Sensitivity to rocuronium-induced neuromuscular block and reversibility with sugammadex in a patient with myotonic dystrophy. Case Rep Anesthesiol. 2012;2012:107952. doi: 10.1155/2012/107952. Epub 2012 Apr 9. PMID 22606401
- [Background] Huang L, Chen D, Li S. Streptozotocin diabetes attenuates the effects of nondepolarizing neuromuscular relaxants on rat muscles. Korean J Physiol Pharmacol. 2014 Dec;18(6):461-7. doi: 10.4196/kjpp.2014.18.6.461. Epub 2014 Dec 30. PMID 25598659